CLINICAL TRIAL: NCT03314116
Title: Assessment of Risk Factors for Hearing Loss as a Result of Exposure to Noise During Military Training in the IDF (Israel Defense Forces), and Examination of the Effectiveness of Hearing Protection Video vs Formal Training.
Brief Title: Risk Factors for Hearing Loss as a Result of Exposure to Noise During Military Training in the IDF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, Sharon Ohayon, Principal Investigator, Medical Corps, Israel Defense Force
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1796-2017
Record Dates: First submitted 2017-09-16; First posted 2017-10-19 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hearing Loss, Noise-Induced
Keywords: hearing loss During basic training, otoacoustic emission
MeSH Terms: conditions — Hearing Loss, Noise-Induced

STUDY DESIGN:
Intervention Model Description: All participants will be randomly assigned to two groups:
  The video group will be guided by a 7-minute video that explains the importance of using ear plugs and correct installation.
  The control group, will be instructed to use earplugs properly, including practical exercises by a medic
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video group (Experimental): guided by a 7-minute video that explains the importance of using ear plugs and correct installation.
  Interventions: Other: Guidance on auditory protection
- control group (No Intervention): instructed to use earplugs properly, including practical exercises by a medic

INTERVENTIONS:
Other: Guidance on auditory protection — by video or medic
  Arms: video group

SUMMARY:
As part of the proposed work, the investigators would like to examine whether there is a need to use a training video to train IDF combat soldiers to improve the use of ear plugs and to prevent hearing loss from exposure to noise, and to characterize the hearing impaired epidemiology of recruits and the basic rate of hearing loss During basic training.

DETAILED DESCRIPTION:
1. Auditory screening examination using an OAE (Oto Acoustic Emission) device during the first week of training in the unit and before starting to be exposed to noise .
2. If the indication obtained by the OAE device is negative, the soldier will be transferred to perform an audiometer test by a medic.
3. If the audiometer is subjected to a significant drop (over 25 decibels), the soldier will be referred to an audiologic examination that includes a comprehensive hearing test and an examination by the ENT (Ear, Nose and Throat).
4. All participants will be randomly assigned to two groups after signing an agreement form:

   A - The video group - will be guided by a screening of a 7 minute video that explains the importance of using ear plugs and correct installation.

   B- The control group, will be instructed to use earplugs properly, including practical exercises by a medic.
5. After two months of training, all participants will undergo further instruction in the use of earplugs, the video clip group and the control group trained by a medic only,
6. Towards the end of the training After six months of the recruitment, the investigators will perform an additional hearing test for all the participants in order to compare the results to the examination performed near their recruitment. Similar to the first stage, the test will be performed using an OAE device.
7. A comparison shall be made in the auditory results data between the group that underwent training via video and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Soldiers who joined the IDF from August 2018

Exclusion Criteria:

* Lack of informed consent.
* recruits who have auditory impairment that is disqualified from fighting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparative impact of military training (infantry, armor and artillery) on hearing loss after full training | 12 months
  The study will measure hearing loss using an Oto Acoustic Emission (OAE) measuring device and an Audiometer test. The results after complete training will be compared against the results obtained prior to training

SECONDARY OUTCOMES:
Percentage of soldiers in combat units which suffer from hearing loss before starting military training | 12 months
Percentage of soldiers in combat units which suffer from hearing loss after completing military training classified to the two groups in the study | 12 months
  The study will investigate the effectiveness of a demonstration video as an audio protection tutorial to prevent hearing loss from exposure to noise in trained fighters. This will be measured against a control group which undergo frontal demonstration by a medic.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Ohayon, MD, Principal Investigator — International Diabetes Federation
Locations (1):
- IDF, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muchnik C, Amir N, Shabtai E, Kaplan-Neeman R. Preferred listening levels of personal listening devices in young teenagers: self reports and physical measurements. Int J Audiol. 2012 Apr;51(4):287-93. doi: 10.3109/14992027.2011.631590. Epub 2011 Nov 28. PMID 22122401
- [Background] Rabinowitz PM, Slade MD, Galusha D, Dixon-Ernst C, Cullen MR. Trends in the prevalence of hearing loss among young adults entering an industrial workforce 1985 to 2004. Ear Hear. 2006 Aug;27(4):369-75. doi: 10.1097/01.aud.0000224125.12338.9a. PMID 16825886
- [Background] Muhr P, Mansson B, Hellstrom PA. A study of hearing changes among military conscripts in the Swedish Army. Int J Audiol. 2006 Apr;45(4):247-51. doi: 10.1080/14992020500190052. PMID 16684706
- [Background] Toh ST, Lu P, Ong M, Seet B. Prevalence of hearing disorders in Singapore military conscripts: a role for routine audiometry screening? Singapore Med J. 2002 Dec;43(12):622-7. PMID 12693766
- [Background] Axelsson A, Rosenhall U, Zachau G. Hearing in 18-year-old Swedish males. Scand Audiol. 1994;23(2):129-34. doi: 10.3109/01050399409047497. PMID 8085113
- [Background] Gold S, Attias J, Cahani M, Shahar A. [Hearing loss as a result of basic military training]. Harefuah. 1989 Apr 2;116(7):377-9. Hebrew. PMID 2737562
- [Background] Ylikoski J. Acute acoustic trauma in Finnish conscripts. Etiological factors and characteristics of hearing impairment. Scand Audiol. 1989;18(3):161-5. doi: 10.3109/01050398909070741. PMID 2814330
- [Background] Murphy WJ, Themann CL, Murata TK. Hearing protector fit testing with off-shore oil-rig inspectors in Louisiana and Texas. Int J Audiol. 2016 Nov;55(11):688-98. doi: 10.1080/14992027.2016.1204470. Epub 2016 Jul 14. PMID 27414471
- [Background] Cassano F, Aloise I, Labianca G, Gaccione V, Mazzotta C, Cardascia F, Garavaglia M, Scarselletta RS, Di Lorenzo L. [Measurement of real personal noise attenuation using earplugs with the E-A-Rfit system]. Med Lav. 2013 May-Jun;104(3):213-23. Italian. PMID 23879065